CLINICAL TRIAL: NCT03656393
Title: Observational Clinical Trial of Adjuvant Chemotherapy for Non-squamous Cell Carcinoma of Non-small Cell Lung Cancer
Brief Title: To Evaluate the Efficacy and Safety of Gefitinib in Adjuvant Chemotherapy for Lung Adenocarcinoma
Acronym: RCTACSCNSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZLY2017024
Record Dates: First submitted 2018-07-17; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: NSCLC; EGFR
Keywords: EGFR; NSCLC; Carboplatin; vinorelbine; Gefitinib
MeSH Terms: interventions — Gefitinib; Vinorelbine; Carboplatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefitinib therapy group (Experimental): Patients are treated with Gefitinib (250 mg, orally, every day) for 56 days and then have an operation. If there is progress after intervention, Patients are further treated with pemetrexe (500 mg/m2, intravenously drip, once a week) plus cisplatin (75 mg/m2, iv. once a week) for 4 weeks.
  Interventions: Drug: Gefitinib
- Vinorelbine combination therapy group (Active Comparator): Patients are treated with vinorelbine (60 mg/m2, orally, Once every three weeks) plus carboplatin (AUC5, intravenously drip, once a week) for 6 weeks and then have an operation. If there is progress after intervention, Patients are further treated with pemetrexe (500 mg/m2, intravenously drip, once a week) plus cisplatin (75 mg/m2, iv. once a week) for 4 weeks.
  Interventions: Drug: Vinorelbine; Drug: Carboplatin

INTERVENTIONS:
Drug: Gefitinib — Gefitinib (250 mg, orally, every day) for 56 days
  Other Names: Iressa
  Arms: Gefitinib therapy group
Drug: Vinorelbine — Vinorelbine (60 mg/m2, orally, Once every three weeks) for 6 weeks
  Other Names: 5'-noranhydrovinblastine; 5-Nonylthio-8-methylthio-chinolin
  Arms: Vinorelbine combination therapy group
Drug: Carboplatin — Carboplatin (AUC5, intravenously drip, once a week) for 6 weeks
  Other Names: Paraplatin; Carboplat; Ercar
  Arms: Vinorelbine combination therapy group

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of targeted gefitinib versus oral vinorelbine and carboplatin in EGFR-mutant NSCLC patients.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of targeted gefitinib versus oral vinorelbine and carboplatin in EGFR-mutant NSCLC patients. The purpose is to explore the role of TKI in neoadjuvant therapy, and to further improve disease-free survival (DFS) and pathologic complete remission (pCR) in EGFR-mutant populations; and reduce surgical complications and mortality.

OBJECTIVES: To evaluate the efficacy of oral gefitinib versus neoadjuvant vinorelbine and carboplatin in operable stage II-IIIA EGFR-mutant non-squamous NSCLC patients, with a 2-year disease-free survival rate. 2yDFS).

Secondary objective: To evaluate pCR, 0RR, and other efficacy measures (safety, complete) for oral gefitinib vs. neoadjuvant vinorelbine and carboplatin in patients with operable stage II-IIIA EGFR-mutant non-squamous cell carcinoma NSCLC. Resection rate, tumor regression, mediastinal lymph node clearance, perioperative complications, and mortality rate).

ELIGIBILITY:
Inclusion Criteria:

1. The pathological diagnosis is non-squamous cell carcinoma and non-small cell lung cancer. The pre-treatment tumor stage is stage II-IIIA;
2. The gene detects EGFR mutations is positive;
3. The age is between 18-70 years;
4. ECOG 0-1;
5. Liver and kidney function and Bone marrow hematopoiesis is normal;
6. There are no serious systemic, respiratory, cardiovascular and other important systemic dysfunctions and severe malnutrition;
7. No other malignant diseases within 5 years;
8. Patients who have not received radiotherapy, systemic chemotherapy, or biological therapy;
9. Understand the whole process of the trial and voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

1. The tumor has invaded the surrounding tissue;
2. Preoperative evidence suggests that distant metastases of the lesion include contralateral mediastinal lymph node metastasis;
3. Arrhythmias require anti-arrhythmia therapy (β-blocker or digoxin Except), symptomatic coronary artery disease or myocardium. Ischemic or congestive heart failure exceeds NYHA class II;
4. severe hypertension with poor drug control;
5. moderate to severe proteinuria;
6. HIV fluHistory of infection or active chronic hepatitis B or C;
7. Malnutrition, decompensation of organ function;
8. History of chest radiotherapy;
9. Incomplete inflammation of eyes;
10. Patients with seizures that need to be treated;
11. Interstitial pneumonia;
12. Drug abuse and others that may interfere with patients' participation in the study or studyThe assessment of the results has an impact;
13. Allergies to the study drug are known or suspected to be allergic to or administered to any drug associated with this test;
14. Any instability. The condition of the patient may jeopardize patient safety and compliance;
15. Pregnancy or breastfeeding women and having fertility without adequate contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
2y DFS | 2 years
  2-year disease-free survival

SECONDARY OUTCOMES:
ORR | 6 months
  objective response rates

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Chen, Doctor, Study Director — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China